CLINICAL TRIAL: NCT06886412
Title: The Effect of Breastfeeding and Maternal Holding on Reducing Pain During Vaccination in Infants
Brief Title: Non-Pharmacological Methods for Reducing Pain During Vaccination in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, Emel AVÇİN, Lecturer Dr, University of Yalova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Emel Avcin Pain
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Pain; Breast Feeding; Maternal Behavior
Keywords: Pain; Vaccines; Nursing; Breastfeeding; Maternal holding; Infants
MeSH Terms: conditions — Pain; Breast Feeding

STUDY DESIGN:
Intervention Model Description: Randomized controlled and quasi-experimental research
Who Masked: Care Provider
Masking Description: During randomization, a separate card color will be assigned for each of the three groups. These cards will be placed inside a black pouch, and the infant's mother will not be able to see them. The card selection will be carried out by a nurse working in the unit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Maternal Holding Group (Experimental): Five minutes before the vaccination procedure, the infant will be handed to the mother in a position suitable for vaccination and will remain in her arms throughout the procedure. It will be checked that the infant's diaper has been changed..The mother will be informed about the importance of stabilizing the leg to be vaccinated during the procedure and will be instructed to hold the infant in a comfortable position. The mother will hold the infant in her lap, using one arm and hand to secure the infant's arms and the other arm and hand to hold the infant's legs. The infant's pain level will be assessed using the Neonatal Infant Pain Scale (NIPS) before, during, and after the vaccination procedure. Crying duration will be measured using a mobile phone stopwatch and recorded in the application record form. The final NIPS assessment and crying duration measurement will be performed 3 minutes after the procedure.
  Interventions: Behavioral: Maternal Holding Intervention Group
- Breast Feeding Group (Experimental): Before the vaccination procedure, the infant and mother will be taken to the vaccination room. The infant's diaper will be checked to ensure it has been changed. The mother will be asked whether the infant has been fed at least 30 minutes before the procedure. The mother will be instructed to sit comfortably on the examination table with her back supported against the wall. The mother will then take the infant in her arms, and the infant will be placed in a cradle hold breastfeeding position. The infant will be handed to the mother 2 minutes before the procedure, and breastfeeding will begin. The infant's pain level will be assessed using the Neonatal Infant Pain Scale (NIPS) before, during, and after the vaccination procedure. Crying duration will be measured using a mobile phone stopwatch and recorded in the application record form. The final NIPS assessment and crying duration measurement will be performed 3 minutes after the procedure.
  Interventions: Behavioral: Breast Feeding Intervention Group
- Control Group (No Intervention): The infants in the control group will receive their vaccinations in the same manner as routine vaccination procedures. Before the vaccination procedure, the infant and their parent will be taken to the room where the procedure will take place, and the infant will be laid on the examination table. During the procedure, the mother will remain next to her infant. To restrict the movement of the infant's legs during the vaccination, the nurse will stabilize the infant's leg with one hand while performing the procedure with the other hand. No non-pharmacological methods will be applied during the procedure. The infant's pain level will be assessed using the Neonatal Infant Pain Scale (NIPS) before, during, and after the vaccination. Crying duration will be measured using a mobile phone stopwatch and recorded in the application record form. The final NIPS assessment and crying duration measurement will be performed 3 minutes after the procedure.

INTERVENTIONS:
Behavioral: Maternal Holding Intervention Group — The infant is required to be held in the mother's arms before, during, and after the procedure. The maternal holding method will be shown or explained to the mother by the researchers.
  Arms: Maternal Holding Group
Behavioral: Breast Feeding Intervention Group — The infant's mother is instructed to begin breastfeeding 2 minutes before the procedure, continuing during and after the procedure. The breastfeeding position for the infant will be shown or explained to the mother by the researchers.
  Arms: Breast Feeding Group

SUMMARY:
Pain management in infants is a medical responsibility of all members of the healthcare team, and nurses hold a privileged role in this regard. The primary goal of pain management is to accurately assess and identify the infant's pain at an early stage, support the development of coping mechanisms through both pharmacological and non-pharmacological methods, and minimize the pain experience as much as possible. Pain management achieved through non-pharmacological interventions constitutes a safe, non-invasive, cost-effective, and independently performed nursing practice. This randomized controlled study was conducted to determine the effect of non-pharmacological methods, specifically maternal holding and breastfeeding, on reducing pain during vaccination in infants.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy,
* Aged between 4 weeks and 6 months,
* Parents have given verbal and written consent to participate in the study,
* Born at term (37 weeks of gestation or later),
* Scheduled for vaccination under the Ministry of Health's vaccination program,
* Not having taken analgesics/antipyretics in the last 4 hours before the procedure,
* Having a normal body temperature (between 36.5°C and 37.1°C).

Exclusion Criteria:

* Having a chronic or mental illness, or a congenital anomaly,
* Being older than 6 months,
* Having a body temperature above 37.1°C,
* Receiving analgesics, sedatives, or any other medication.

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2025-02-02 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Evaluation of pain and crying duration in the infant held in the mother's arms during the vaccination procedure | Two minutes before the procedure, during the procedure, and three minutes after the procedure.
  The pain of the infant held in the mother's arms will be measured using the Neonatal Infant Pain Scale 2 minutes before the procedure, during the procedure, and 3 minutes after the procedure. The crying duration before and after the procedure will be measured using a stopwatch.
Evaluation of pain and crying duration in the infant held in the breast feeding during the vaccination procedure | Two minutes before the procedure, during the procedure, and three minutes after the procedure.
  The pain of the infant using the breastfeeding method will be measured using the Neonatal Infant Pain Scale 2 minutes before the procedure, during the procedure, and 2 minutes after the procedure. The crying duration before and after the procedure will be measured using a stopwatch.

CONTACTS AND LOCATIONS:
Overall Officials: EMEL AVÇİN, Doctor, Principal Investigator — University of Yalova
Locations (1):
- Yalova University, Yalova, Turkey (Türkiye)